CLINICAL TRIAL: NCT06247982
Title: Bail-Out Stenting and Target-vessel Failure After Drug Coated Balloon Coronary percutaneouS Angioplasty for de Novo Lesions: the BOSS Study
Brief Title: Bail-Out Stenting and Target-vessel Failure After Drug Coated Balloon Coronary percutaneouS Angioplasty for de Novo Lesions
Acronym: BOSS
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: BOSS study
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: DCB; De Novo Stenosis; PCI
Keywords: DCB; PCI; de novo; Bail-out stenting; TVF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DCB de novo PCI: All patients who received a de novo DCB PCI
- BOS PCI: All patients who received a stent after DCB treatment of de novo coronary lesion because of high grade dissection or recoil more than 30%

SUMMARY:
The goal of this observational retrospective and prospective multicentric trial is to learn about the impact of bail-out stenting (BOS) after drug coated balloon (DCB) percutaneous coronary angioplasty (PCI) in de novo coronary stenosis.The main question to answer is:

- if BOS PCI leads to an higher rate of 1-year target vessel failure that DCB-only PCI.

Participants will receive DCB PCI in de novo coronary stenosis. Treatments they'll be given should be:

* DCB-only PCI
* BOS PCI

Researchers will compare DCB-only and BOS group to see if addictive stent implantation for DCB-PCI complication is relate to an higher rate of target vessel failure.

Target vessel is the primary endpoint, defined as:

* cardiovascular death
* target vessel myocardial infarction
* clinical driven target vessel revascularization
* angiographic restenosis

DETAILED DESCRIPTION:
Drug coated balloon (DCB) percutaneous coronary intervention (PCI) has been shown to be as effective as last generation drug eluting stent (DES) PCI in many randomized trials. However a not negligible rate of patients must receive a bail-out stenting (BOS) implantation after DCB-PCI. Only some studies report that the rate of MACE of these patients is higher than DCB-only or DES-PCI ones. Even if the BOS patients MACE rate is two times more than DCB-only or DES-only, due to the small amount of BOS patients in these studies there were not a statistically significant difference.

According to these evidence, BOSS study researchers will compare target vessel failure (TVF) rate in DCB-only and BOS group resulting from all vessel size de novo coronary artery stenosis DCB-PCI.

TVF as primary endpoint will include:

* cardiovascular death
* target vessel myocardial infarction (TV-MI). According to the third universal definition of myocardial infarction TV-MI will be considered a non fatal myocardial infarction with the evidence of myocardial necrosis in the vascular territory of previously treated target vessel
* clinical driven target vessel revascularization (CD-TVR). CD-TVR will be considered as any repeat intervention of any segment of the target vessel, defined as the entire major coronary vessel proximal and distal to the target lesion.
* Angiographic restenosis. It will considered in case of restenosis as either a > 50% loss of initial gain of the target lesion.

The trial will enroll all patients who received a de novo DCB-PCI from January 2020 to December 2023. The population will be divided into two groups:

* DCB-only PCI
* BOS PCI

Bail-out stenting will be done in case of high grade coronary dissection (> or equal to NHLBI grade C) or in case of > 30% recoil, according with International DCB Consensus.

ELIGIBILITY:
Inclusion Criteria:

* De novo DCB PCI of at least one coronary artery
* Hybrid PCI of bifurcation (main branch stent and side branch DCB)
* Hybrid PCI of coronary artery with more than one stenosis (at least 10 mm of distance between edge of stent and DCB PCI segment)

Exclusion Criteria:

* in-stent restenosis
* more than 1 year life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All de novo DCB PCI ≥ 18 years-old patients who meet inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-01-28 (Estimated)

PRIMARY OUTCOMES:
Target Vessel Failure of de novo PCI | 1 year
  Number of patients with the composite endpoint (number of cardiovascular death, TV-MI, CD-TVR, angiographic restenosis)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Ghetti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico di Sant'Orsola
Locations (1):
- Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No